CLINICAL TRIAL: NCT00573443
Title: A Double-Blind, Randomized, Placebo-Controlled, Multicenter Study to Assess the Safety and Efficacy and to Determine the Pharmacokinetics of Two Doses of AVP-923 (Dextromethorphan/Quinidine) in the Treatment of Pseudobulbar Affect (PBA) in Patients With Amyotrophic Lateral Sclerosis (ALS) and Multiple Sclerosis (MS)
Brief Title: Safety and Efficacy of AVP-923 in PBA Patients With ALS or MS
Acronym: STAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Avanir Pharmaceuticals (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-AVR-123
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Results first posted 2013-07-10 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Pseudobulbar Affect (PBA)
Keywords: Amyotrophic Lateral Sclerosis (Lou Gehrig's disease, ALS); Multiple Sclerosis (MS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Multiple Sclerosis | interventions — Dextromethorphan; Quinidine; dextromethorphan - quinidine combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DM 30 mg/Q 10 mg (Experimental): AVP-923-30/10 Capsules (30 mg dextromethorphan/10 mg quinidine)administered once daily for 1 week and then twice daily for 11 weeks
  Interventions: Drug: dextromethorphan hydrobromide 30 mg and quinidine sulfate 10 mg
- DM 20 mg/ Q 10 mg (Experimental): AVP-923-20/10 Capsules (20 mg dextromethorphan/10 mg quinidine)administered once daily for 1 week and then twice daily for 11 weeks
  Interventions: Drug: dextromethorphan hydrobromide 20 mg and quinidine sulfate 10 mg
- Placebo (Placebo Comparator): Placebo Capsules once daily for 1 week and then twice daily for an additional 11 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: dextromethorphan hydrobromide 20 mg and quinidine sulfate 10 mg — Dextromethorphan hydrobromide (DM) and quinidine sulfate (Q) capsules (AVP-923 capsules), containing DM 20 mg/ Q 10 mg, taken once daily for 1 week and then twice daily for 11 consecutive weeks to complete a 12-week period
  Other Names: AVP-923; Nuedexta™; DM 20 mg/ Q 10 mg; DMQ
  Arms: DM 20 mg/ Q 10 mg
Drug: dextromethorphan hydrobromide 30 mg and quinidine sulfate 10 mg — Dextromethorphan hydrobromide (DM) and quinidine sulfate (Q) capsules (AVP-923 capsules), containing DM 30 mg/ Q 10 mg taken once daily for 1 week and then twice daily for 11 consecutive weeks to complete a 12-week period
  Other Names: AVP-923; DM 30 mg/ Q 10 mg; DMQ
  Arms: DM 30 mg/Q 10 mg
Drug: Placebo — Placebo capsules (identical in appearance to AVP-923 capsules being studied in this trial), taken once daily for 1 week and then twice daily for 11 consecutive weeks to complete a 12-week period
  Arms: Placebo

SUMMARY:
Objectives of the study are to evaluate the safety, tolerability, and efficacy of two different doses of AVP-923 (capsules containing either 30 mg of dextromethorphan hydrobromide and 10 mg of quinidine sulfate [AVP-923-30] or 20 mg of dextromethorphan hydrobromide and 10 mg of quinidine sulfate [AVP-923-20]) when compared to placebo, for the treatment of PBA in a population of patients with amyotrophic lateral sclerosis (ALS) or multiple sclerosis (MS) over a 12-week period. An additional objective is to determine the pharmacokinetic parameters of the two different doses of AVP-923 in a subset of the study population.

Pseudobulbar Affect (PBA) is a condition characterized by involuntary, sudden and frequent episodes of laughing and/or crying out of proportion or incongruous to the underlying emotion of happiness or sadness Other terms used to describe this condition include emotional lability, emotionalism, emotional incontinence, emotional discontrol, excessive emotionalism, and pathological laughing and crying. The outbursts can occur spontaneously or in response to provocative stimuli such as questions or events.

A body of evidence suggests that PBA can be modulated through pharmacologic intervention.

Dextromethorphan (DM) is a low-affinity uncompetitive antagonist of the N-Methyl-D-aspartate (NMDA) receptor, reducing the level of excitatory activity. DM also acts at the phencyclidine-binding site, which is part of the NMDA receptor complex. DM is a sigma receptor agonist, suppressing the release of excitatory neurotransmitters.

Quinidine (Q) is a known potent inhibitor of cytochrome P450 2D6 (CYP2D6), that decreases the metabolism of dextromethorphan and helps to achieve sustained and therapeutic levels of this drug.

ELIGIBILITY:
Main Inclusion Criteria:

* The patient has a diagnosis of Amyotrophic Lateral Sclerosis (according to El Escorial Criteria, WFN, 1998) and the time from diagnosis of ALS is not be longer than 30 months, or the patient has a diagnosis of multiple sclerosis or probable multiple sclerosis (according to McDonald criteria, 2001)
* The patient has a clinical history and clinical relevant symptoms of Pseudobulbar Affect (PBA)
* CNS-LS score at baseline is 13 or greater

Main Exclusion Criteria:

* Patients with myasthenia gravis
* Any personal history of complete heart block, QTc prolongation, or torsades de pointes
* Any family history of congenital QT interval prolongation syndrome
* Patients with known sensitivity to quinidine, dextromethorphan or opiate drugs (codeine, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2007-12; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Hepner, M.D., Study Director — Avanir Pharmaceuticals
Locations (62):
- United States (45):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Neuromuscular Research Center, Scottsdale, Arizona
  - South Coast Clinical Trials, Anaheim, California
  - UCI Medical Center, Irvine, California
  - Center for Neurologic Study, La Jolla, California
  - UCLA School of Medicine, Los Angeles, California
  - The Forbes Norris MDA/ALS Research Center - California Pacific Medical Center, San Francisco, California
  - The ALS Center at UCSF, San Francisco, California
  - University of Colorado at Denver & Health Science Center, Aurora, Colorado
  - Neuroscience Center, Fort Lauderdale, Florida
  - Mayo Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Suncoast Neuroscience Associates, St. Petersburg, Florida
  - The ALS Center at Emory University, Atlanta, Georgia
  - Neurology Specialists of Decatur of Decatur, Decatur, Georgia
  - Northwestern University, Chicago, Illinois
  - Consultants in Neurology, Northbrook, Illinois
  - University of Kentucky Health Care - Dept. of Neurology, Lexington, Kentucky
  - The John Hopkins Universitiy, Baltimore, Maryland
  - Massachusets General Hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - St.Louis University - Neuromuscular Clinic, St Louis, Missouri
  - Advanced Neurology Specialists, Great Falls, Montana
  - Neurology Associates, Lincoln, Nebraska
  - Universitiy of Nevada, Las Vegas, Nevada
  - Upstate Clinical Research, Albany, New York
  - Jacobs Neurological Institute, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - Neurological Institute - Columbia Presbyterian Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke Universitiy Medical Center, Durham, North Carolina
  - Department of Neurology - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State Universitiy, Columbus, Ohio
  - Oregon Health Science University, Portland, Oregon
  - Drexel University - Department of Neurology, Philadelphia, Pennsylvania
  - The ALS Center - Penn Neurological Institute - The University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - The Methodist Hospital - Baylor College of Medicine, Houston, Texas
  - Department of Neuropsychiatry - Texas Tech University, Lubbock, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - Universitiy of Vermont, Burlington, Vermont
  - West Virginia University, Morgantown, West Virginia
  - Dean Foundation, Madison, Wisconsin
- Argentina (11):
  - FACENE, Buenos Aires, Buenos Aires F.D.
  - IADIN, Buenos Aires, Buenos Aires F.D.
  - Hospital Italiano, Buenos Aires, Buenos Aires F.D.
  - INEBA, Buenos Aires, Buenos Aires F.D.
  - Hospital Ramos Mejia, Buenos Aires, Buenos Aires F.D.
  - Hospital Britanico, Buenos Aires, Buenos Aires F.D.
  - Policlinico Bancario, Buenos Aires, Buenos Aires F.D.
  - FLENI, Buenos Aires, Buenos Aires F.D.
  - Hospital Militar Regional de Cordoba, Córdoba, Córdoba Province
  - Instituto Medico Rodriguez Alfici, Godoy Cruz, Mendoza Province
  - Instituto de Neurociencias Rosario, Rosario, Santa Fe Province
- Brazil (6):
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte, M G
  - Hospital de Clínicas-UFPR, Curitiba, Paraná
  - Hospital da Restauração, Recife, Pernambuco
  - Hospital Universitário Clementino Fraga Filho, Rio de Janeiro, Rio de Janeiro
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital das Clínicas da Faculdade de Medicina da Universidade São Paulo, São Paulo, São Paulo

REFERENCES:
- [Result] Pioro EP, Brooks BR, Cummings J, Schiffer R, Thisted RA, Wynn D, Hepner A, Kaye R; Safety, Tolerability, and Efficacy Results Trial of AVP-923 in PBA Investigators. Dextromethorphan plus ultra low-dose quinidine reduces pseudobulbar affect. Ann Neurol. 2010 Nov;68(5):693-702. doi: 10.1002/ana.22093. PMID 20839238

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects diagnosed with pseudobulbar affect (PBA) secondary to amyotrophic lateral sclerosis (ALS) or multiple sclerosis (MS).
Groups:
- AVP-923-30: AVP-923 capsules containing 30 mg dextromethorphan (DM) and 10 mg quinidine (Q) taken orally once daily for 1 week and twice daily for 11 additional consecutive weeks for a 12 week double-blind (DB) period. Subjects who completed the DB period of this treatment arm could begin an optional 12 week open-label extension (OLE) period taking AVP-923 capsule containing 30 mg DM and 10 mg Q twice daily.
- AVP-923-20: AVP-923 capsules containing 20 mg DM and 10 mg Q taken orally once daily for 1 week and twice daily for 11 additional consecutive weeks for a 12 week DB period. Subjects who completed the DB period of this treatment arm could begin an optional 12 week OLE period taking AVP-923 capsule containing 30 mg DM and 10 mg Q twice daily.
- Placebo: Capsules containing placebo once daily for 1 week and twice daily for 11 additional consecutive weeks for a 12 week DB period. Subjects who completed the DB period of this treatment arm could begin an optional 12 week OLE period taking AVP-923 capsule containing 30 mg DM and 10 mg Q twice daily.
Period: Double-Blind Phase
Arm/Group | AVP-923-30 | AVP-923-20 | Placebo
Started | 110 | 107 | 109
Subjects With PBA Secondary to ALS | 65 | 68 | 64
Subjects With PBA Secondary to MS | 45 | 39 | 45
Completed | 101 | 88 | 94
Not Completed | 9 | 19 | 15
Not completed — Lost to Follow-up | 1 | 3 | 2
Not completed — Exacerbation of MS symptoms | 1 | 0 | 1
Not completed — Adverse Event | 1 | 5 | 0
Not completed — Serious Adverse Event (AE) | 2 | 3 | 1
Not completed — Medication refusal due to AE | 2 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 7
Not completed — Protocol Violation | 0 | 2 | 1
Not completed — Other | 0 | 2 | 3
Period: Open-Label Extension Phase
Arm/Group | AVP-923-30 | AVP-923-20 | Placebo
Started | 253 (Subjects who completed any of the arms in the DB phase had the option to enroll in this OLE phase) | 0 (DB period of this arm could begin an optional 12 week OLE period taking AVP-923-30.) | 0 (DB period of this arm could begin an optional 12 week OLE period taking AVP-923-30.)
Subjects With PBA Secondary to ALS | 146 | 0 (DB period of this arm could begin an optional 12 week OLE period taking AVP-923-30.) | 0 (DB period of this arm could begin an optional 12 week OLE period taking AVP-923-30.)
Subjects With PBA Secondary to MS | 107 | 0 (DB period of this arm could begin an optional 12 week OLE period taking AVP-923-30.) | 0 (DB period of this arm could begin an optional 12 week OLE period taking AVP-923-30.)
Completed | 235 | 0 (DB period of this arm could begin an optional 12 week OLE period taking AVP-923-30.) | 0 (DB period of this arm could begin an optional 12 week OLE period taking AVP-923-30.)
Not Completed | 18 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Exacerbation of MS symptoms | 2 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Serious Adverse Event | 5 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Other | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AVP-923-30 | AVP-923-20 | Placebo | Total
Number analyzed (Participants) | 110 | 107 | 109 | 326
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.08 (11.016) | 50.81 (11.114) | 50.27 (11.939) | 51.39 (11.356)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 54 | 59 | 177
  Male | 46 | 53 | 50 | 149

OUTCOME MEASURES:

1. Primary Outcome: PBA Episode Rate Ratio (Post/Pre), Regression Adjusted
Description: Episodes were counted each day and recorded in a daily diary. The outcome measure is the ratio of the episode rate over the 84-day treatment period to the rate during the baseline period, adjusted for study site, and underlying disease using longitudinal negative binomial regression.
Time Frame: Baseline to Day 84
Population: Intent-to-Treat (ITT) population - included all randomized subjects for the double-blind phase and all enrolled subjects for the open-label extension phase.
Measure: Least Squares Mean (95% Confidence Interval); unit: Unit-free (ratio of episodes/week)
Arm/Group | AVP-923-30 | AVP-923-20 | Placebo
Number analyzed (Participants) | 110 | 107 | 109
Unit-free (ratio of episodes/week) | 0.247 (3.447) [0.233 to 0.262] | 0.237 (6.048) [0.224 to 0.251] | 0.465 (6.642) [0.441 to 0.489]
Statistical Analysis 1: Comparison: AVP-923-30 vs Placebo; Analysis of PBA episode rates used longitudinal negative binomial regression with treatment, period, diagnosis and study site to estimate pre-post changes in log mean episode rate for each treatment group. Null hypothesis of equal pre-post episode rate reductions were tested: AVP-923-30/placebo = 1; Test type: Superiority or Other; p < 0.0001, Regression, Longitudinal neg. binomial; Ratio of episode-rate reduction ratios = 0.5312, 95% CI 2-sided [0.4939 to 0.5714]
Statistical Analysis 2: Comparison: AVP-923-20 vs Placebo; Analysis of PBA episode rates used longitudinal negative binomial regression with treatment, period, diagnosis and study site to estimate pre-post changes in log mean episode rate for each treatment group. Null hypothesis of equal pre-post episode rate reductions were tested: AVP-923-20/placebo = 1; Test type: Superiority or Other; p < 0.0001, Regression, Longitudinal neg. binomial; Ratio of episode-rate reduction ratios = 0.5103, 95% CI 2-sided [0.4755 to 0.5477]

2. Secondary Outcome: Mean Change From Baseline in CNS-LS Total Score by Visit
Description: Center for Neurologic Studies-Lability Scale (CNS-LS) is an instrument for the measurement of PBA that has been validated for the use in patients with ALS and MS. It is a 7-item self-report questionnaire that measures the frequency and severity of PBA episodes, including assessments of labile laughter and labile tearfulness,and provides a score for total PBA (total score can range from 7-35). The following 5-point scoring was used: 1=Applies never, 2=Applies rarely, 3=Applies occasionally, 4=Applies frequently, 5=Applies most of the time. A score of 13 or higher may suggest PBA, and the higher the score the more severe the episodes.
Time Frame: Baseline, Day 15, Day 29, Day 57, Day 84
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | AVP-923-30 | AVP-923-20 | Placebo
Number analyzed (Participants) | 110 | 107 | 109
Scores on a Scale
  Day 15 (Visit2) | -6.77 (5.239) | -6.27 (5.552) | -4.58 (4.982)
  Day 29 (Visit 3) | -8.03 (5.591) | -7.62 (5.421) | -5.70 (5.034)
  Day 57 (Visit 4) | -8.59 (5.745) | -8.89 (5.501) | -5.66 (5.038)
  Day 84 (Visit 5) | -8.17 (6.104) | -8.24 (6.126) | -5.72 (5.280)

3. Secondary Outcome: Mean Change From Baseline to Day 84 in Neuropsychiatric Inventory (NPI-Q) Frequency and Severity Score (EE Population)
Description: The NPI is a retrospective (to 1 month) caregiver-informant interview assessing frequency and severity of 12 neuropsychiatric symptom domains. The NPI score is based on the sum of the severity ratings (0=absent, 1=mild, 3=severe). The 12 symptom domains include delusions, hallucinations, agitation/aggression, dysphoria/depression, anxiety, euphoria/elation, apathy/indifference, disinhibition, irritability/lability, aberrant motor behaviors, nighttime behavioral disturbances, and appetite/eating abnormalities. The NPI severity score is based on severity ratings (0=absent, 1=mild to 3=severe).
Time Frame: Baseline to Day 84
Population: Efficacy Evaluable (EE) Population - included all subjects who were protocol adherent, defined as those who completed the Day 84 visit or the end-of-study visit within 48 hours of a discontinuation, and who took as least 80% of their scheduled doses prior to discontinuation of the study medication.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | AVP-923-30 | AVP-923-20 | Placebo
Number analyzed (Participants) | 105 | 90 | 98
Scores on a Scale
  Frequency Score | -1.68 (4.102) | -3.09 (6.241) | -1.25 (4.860)
  Severity Score | -0.80 (3.109) | -1.81 (4.206) | -0.91 (4.026)

4. Secondary Outcome: Mean Change From Baseline to Day 84 in Neuropsychiatric Inventory (NPI-Q) Frequency and Severity Score (ITT Population)
Description: as for outcome 3
Time Frame: Baseline to Day 84
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | AVP-923-30 | AVP-923-20 | Placebo
Number analyzed (Participants) | 110 | 107 | 109
Scores on a Scale
  Frequency Score | -1.62 (4.110) | -2.56 (6.205) | -1.33 (4.837)
  Severity Score | -0.74 (3.102) | -1.59 (4.128) | -0.98 (4.008)

5. Secondary Outcome: Mean Change From Baseline at Day 84 in SF-36 (Short-Form) Health Survey Medical Outcome Score by Category
Description: The SF-36 is designed to examine a person's perceived health status. The SF-36 includes one multi-item scale measuring eight health concepts: vitality, physical functioning, bodily pain, general health perceptions, physical role-, emotional role-, social role functioning, and mental health. Answers to each question are scored and summed to produce raw scale scores for each health concept which are then transformed to a 0 - 100 scale, a high score defining a more favorable health state. An aggregate summary measure is calculated by averaging the scores from the eight health concepts.
Time Frame: Baseline and Day 84
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | AVP-923-30 | AVP-923-20 | Placebo
Number analyzed (Participants) | 110 | 107 | 109
Scores on a Scale
  Physical Functioning Scale | -0.90 (17.336) | -5.30 (15.652) | -4.05 (16.381)
  Role Physical Scale | 3.47 (36.747) | -4.26 (39.764) | -1.75 (40.084)
  Bodily Pain Scale | 4.09 (20.861) | 5.84 (20.437) | -1.13 (21.782)
  General Health Scale | -1.47 (17.273) | -2.95 (16.266) | -1.28 (15.824)
  Vitality Scale | -0.90 (17.336) | -5.30 (15.652) | -4.05 (16.381)
  Social Functioning Scale | 9.34 (25.105) | 1.42 (28.577) | -3.09 (28.908)
  Role Emotional Scale | 11.55 (47.711) | -1.81 (45.924) | 2.36 (45.984)
  Mental Health Scale | 5.53 (17.067) | 3.09 (16.877) | -0.28 (13.720)

6. Secondary Outcome: Mean Change From Baseline at Day 84 in Beck Depression Inventory (BDI-II) Total Score
Description: The BDI-II is a 21-item self report instrument intended to assess the existence and severity of symptoms of depression, summed to give a single score. The BDI-II uses a 4-point for each item ranging from 0 to 3. A total score of 0-13 is considered minimal range, 14 to 19 is mild, 20 to 28 is moderate, and 29 to 63 is severe.
Time Frame: Baseline and Day 84
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | AVP-923-30 | AVP-923-20 | Placebo
Number analyzed (Participants) | 110 | 107 | 109
Scores on a Scale | -1.59 (5.294) | -1.03 (5.183) | -0.02 (6.320)

7. Secondary Outcome: Mean Change From Baseline to Day 84 in Pain Rating Scale (PRS) of MS Subjects
Description: Subjects with MS were instructed to also record daily the pain they experienced using the PRS. After evaluating the subject's ability to comply with these requirements, the investigator determined if a caregiver should complete the study diary and assessments. Subjects rated their pain over the past 12 hours on a scale of 0 to 10 (0=none, 10=worst pain ever experienced).
Time Frame: Baseline, Day 15, Day 29, Day 57, Day 84
Population: ITT Population - MS Subjects only
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | AVP-923-30 | AVP-923-20 | Placebo
Number analyzed (Participants) | 45 | 39 | 45
Scores on a Scale | -1.0 (2.39) | -0.7 (1.84) | -0.4 (2.61)

ADVERSE EVENTS:
Groups:
- AVP-923-30 (Double-blind): AVP-923 capsules containing 30 mg dextromethorphan (DM) and 10 mg quinidine (Q) taken orally once daily for 1 week and twice daily for 11 additional consecutive weeks for a 12 week double-blind (DB) period.
- AVP-923-20 (Double-blind): AVP-923 capsules containing 20 mg DM and 10 mg Q taken orally once daily for 1 week and twice daily for 11 additional consecutive weeks for a 12 week DB period.
- Placebo (Double-blind): Capsules containing placebo once daily for 1 week and twice daily for 11 additional consecutive weeks for a 12 week DB period.
- AVP-923-30 (Open Label): Optional 12-week Open Label phase for subjects who completed 12-week DB phase.
Arm/Group | AVP-923-30 (Double-blind) | AVP-923-20 (Double-blind) | Placebo (Double-blind) | AVP-923-30 (Open Label)
Serious Adverse Events (participants affected / at risk) | 8/110 | 9/107 | 10/109 | 14/253
Other Adverse Events (participants affected / at risk) | 66/110 | 65/107 | 63/109 | 123/253
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AVP-923-30 (Double-blind) (N=110) | AVP-923-20 (Double-blind) (N=107) | Placebo (Double-blind) (N=109) | AVP-923-30 (Open Label) (N=253)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 2
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
RESPIRATORY DEPRESSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
INCREASED BRONCHIAL SECRETION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
DYSPHAGIA (Gastrointestinal disorders) | 1 | 0 | 2 | 1
STRIDOR (Gastrointestinal disorders) | 0 | 0 | 0 | 1
RESPIRATORY DISORDER (Gastrointestinal disorders) | 0 | 0 | 0 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 0 | 1 | 0
SYNCOPE (Nervous system disorders) | 1 | 0 | 0 | 0
MUSCLE SPASTICITY (Nervous system disorders) | 0 | 1 | 0 | 0
MULTIPLE SCLEROSIS (Nervous system disorders) | 1 | 0 | 0 | 0
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 0 | 0 | 0 | 2
UROSEPSIS (Infections and infestations) | 0 | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 0 | 0 | 0
INFECTION (Infections and infestations) | 0 | 1 | 0 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 1 | 0
CATHETER RELATED INFECTION (Infections and infestations) | 0 | 1 | 0 | 0
TOOTH INFECTION (Infections and infestations) | 0 | 0 | 0 | 1
SKIN INFECTION (Infections and infestations) | 0 | 0 | 0 | 1
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 | 0 | 0 | 1
APPENDICITIS (Infections and infestations) | 0 | 0 | 0 | 1
POSTOPERATIVE RESPIRATORY DISTRESS (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
FEEDING TUBE COMPLICATION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
COMPLICATION OF DEVICE INSERTION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 2 | 0
SUICIDE ATTEMPT (Psychiatric disorders) | 0 | 1 | 0 | 0
ANXIETY (Psychiatric disorders) | 1 | 0 | 0 | 0
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 | 0 | 0 | 1
OXYGEN SATURATION DECREASED (Investigations) | 0 | 1 | 0 | 0
CARDIAC ENZYMES INCREASED (Investigations) | 0 | 1 | 0 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 0 | 1 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 0 | 1 | 0
DISEASE PROGRESSION (General disorders) | 0 | 1 | 1 | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AVP-923-30 (Double-blind) (N=110) | AVP-923-20 (Double-blind) (N=107) | Placebo (Double-blind) (N=109) | AVP-923-30 (Open Label) (N=253)
NAUSEA (Gastrointestinal disorders) | 14 | 8 | 10 | 15
DIARRHOEA (Gastrointestinal disorders) | 11 | 14 | 7 | 0
CONSTIPATION (Gastrointestinal disorders) | 7 | 6 | 9 | 17
DYSPHAGIA (Gastrointestinal disorders) | 4 | 6 | 2 | 0
DRY MOUTH (Gastrointestinal disorders) | 7 | 2 | 0 | 0
FATIGUE (General disorders) | 9 | 11 | 10 | 30
NASOPHARYNGITIS (Infections and infestations) | 9 | 6 | 8 | 14
URINARY TRACT INFECTION (Infections and infestations) | 8 | 4 | 3 | 19
FALL (Injury, poisoning and procedural complications) | 22 | 14 | 22 | 40
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 7 | 3 | 10 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 | 2 | 8 | 14
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 6 | 5 | 4 | 17
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 16
HEADACHE (Nervous system disorders) | 15 | 15 | 17 | 27
DIZZINESS (Nervous system disorders) | 20 | 11 | 6 | 17
SOMNOLENCE (Nervous system disorders) | 11 | 9 | 10 | 16
DEPRESSION (Psychiatric disorders) | 0 | 1 | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less